CLINICAL TRIAL: NCT01419015
Title: A Clinical Trial of a 20mm Transcatheter Bioprosthetic Valve for Patients With Aortic Stenosis
Brief Title: PREVAIL-20J - Transfemoral Placement of 20mm Aortic Balloon Expandable Transcatheter Valve Trial
Acronym: PREVAIL-20J
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EW-P-002
Record Dates: First submitted 2011-08-16; First posted 2011-08-17 (Estimated); Results first posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Aortic Valve Stenosis
Keywords: SAPIEN XT Valve (20mm); Cardiovascular Disease; Valvular Heart Disease; Aortic Stenosis; Heart Valve Therapy; Transcatheter; Transfemoral; Efficacy endpoints; Indexed Aortic Valve Area; NYHA
MeSH Terms: conditions — Aortic Valve Stenosis; Cardiovascular Diseases; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- TAVI-TF Approach (Experimental): Transcatheter aortic valve implantation and transfemoral approach. SAPIEN XT NovaFlex delivery system will be used.
  Interventions: Device: SAPIEN XT NovaFlex delivery system

INTERVENTIONS:
Device: SAPIEN XT NovaFlex delivery system — Transcatheter aortic valve implantation via transfemoral approach.
  Other Names: SAPIEN XT; NovaFlex delivery system

SUMMARY:
A single arm, prospective multicenter non-randomized pivotal clinical trial evaluating the 20mm Edwards SAPIEN XT™ transcatheter heart valve (model 9300TFX), NovaFlex™ transfemoral delivery system, and crimper accessories. The trial includes a premarket pivotal cohort to evaluate the system performance as well as a post market clinical follow-up phase involving long term follow-up of all patients to evaluate the safety of investigational devices up to 5 years.

DETAILED DESCRIPTION:
Purpose: To evaluate the safety and efficacy of THV-9300 (20mm) for patients who have severe symptomatic aortic stenosis attributed to calcification and degeneration of a valve leaflet and for whom undergoing a surgery safely would be difficult.

Enrollment: 15 patients (No.of patients needed: 12)

Follow-up: Subject data collection will include clinical information at baseline and during the index procedure. Subjects will undergo clinical follow-up at discharge, 30 days, 6 months and annually for 5 years.

Clinical sites:

1)Osaka University Hospital, 2)Kurashiki Central Hospital, 3)Sakakibara Heart Institute, 4) Kokura Memorial Hospital

ELIGIBILITY:
Inclusion Criteria:

* Patients who were judged difficult to safely undergo AVR
* Severe senile degenerative aortic valve stenosis
* NYHA Functional Class II or greater
* Signed Informed Consent

Exclusion Criteria:

* Aortic valve is congenital unicuspid or bicuspid
* Annulus size between < 16 mm or > 19 mm
* LVEF < 20 %

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morimasa Takayama, MD, Principal Investigator — Sakakibara Heart Institute
Locations (4):
- Japan (4):
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - Osaka University Hospital, Suita, Osaka
  - Sakakibara Heart Institute, Fuchū, Toyko

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- 20-mm TF-TAVR: Patients with symptomatic severe aortic stenosis received a 20 mm SAPIEN XT valve through the transfemoral procedure.
Period: Overall Study
Arm/Group | 20-mm TF-TAVR
Started | 17
Completed | 15
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | 20-mm TF-TAVR
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 82.2 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 0
NYHA Class III/IV [Count of Participants; unit: Participants] | 11
Porcelain Aorta [Count of Participants; unit: Participants] | 3
Diabetes [Count of Participants; unit: Participants] | 6
Arrhythmia [Count of Participants; unit: Participants] | 4

OUTCOME MEASURES:

1. Primary Outcome: NYHA Improvement and AVA >= 0.65 cm2
Description: Improvement of the aortic valve area (AVA) and New York Heart Association (NYHA) functional classification from baseline to 1 year after the procedure. NYHA functional classification of heart failure based on how much a patient is limited during physical activity. The rating ranges from I-IV, with the lowest (I) as no limitations and the highest (IV) unable to carry on any physical activity without discomfort. The AVA at 1 year >= 0.65 cm2 indicates improvement. This outcome measure shows the percentage of patients that had an improvement in both NYHA Class and AVA. Note: One patient did not complete a 6-month echo.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | TAVI-TF Approach
Number analyzed (Participants) | 16
Participants | 14

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | TAVI-TF Approach
All-Cause Mortality (participants affected / at risk) | 2/17
Serious Adverse Events (participants affected / at risk) | 8/17
Other Adverse Events (participants affected / at risk) | 11/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAVI-TF Approach (N=17)
Hemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Acute myocardial Infraction (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 1 (1)
Device malposition (General disorders) | 1 (1)
Aortic injury (Injury, poisoning and procedural complications) | 1 (1)
Femoral fracture (Injury, poisoning and procedural complications) | 1 (1)
Cardiac perforation (Injury, poisoning and procedural complications) | 1 (1)
Spinal Compression Fracture (Nervous system disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Cardiac Failure (Cardiac disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAVI-TF Approach (N=17)
Pneumonia (Infections and infestations) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (6)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Cerebral Infraction (Nervous system disorders) | 1 (1)
Dementia (Nervous system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Aortic regurgitation (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Gingival bleeding (Vascular disorders) | 1 (1)
Peripheral ischemia (Vascular disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lower gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Subcutaneous hemorrhage (Skin and subcutaneous tissue disorders) | 1 (1)
Increased Intraocular pressure (Investigations) | 1 (1)
Cataract surgery (Surgical and medical procedures) | 1 (1)
Epidermal necrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Left Leg Block (General disorders) | 1 (1)
Ventricular Extrasystole (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No